CLINICAL TRIAL: NCT04617379
Title: Stretching Exercises and Musculoskeletal Pain Among Employees Working in the Echocardiographic, Ultrasound and Interventional Laboratories
Brief Title: Stretching and Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-003714
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment Group (Experimental): 15 minutes daily stretch for 1 year
  Interventions: Behavioral: Stretching
- Control Group (No Intervention): No stretches

INTERVENTIONS:
Behavioral: Stretching — One-year stretching program for 15 minutes every day
  Arms: Active Treatment Group

SUMMARY:
The purpose of this study is to assess whether a daily, 15-minute stretching routine for one year reduces musculoskeletal pain and improves quality of life in personnel working in the radiology and cardiology departments at Mayo Clinics and Mayo Clinic Health System sites.

ELIGIBILITY:
Inclusion Criteria:

* A 15-minute daily stretching program will be implemented for 1 year.
* Personnel working in the departments of Cardiology and Radiology at Mayo Rochester, - Mayo Scottsdale, and Mayo Jacksonville and Mayo Clinic Health System.
* Willing to complete standardized questionnaires (DASH, ODI) to assess work-related pain at baseline and at 1 year.
* Employees who respond to questionnaires at baseline and 1 year but don't participate in the stretching exercises will be controls for the study.
* Willing and able to provide written, informed consent.

Exclusion Criteria:

* Pregnancy.
* Inability to participate in the stretching exercises for any reason.
* Preexisting musculoskeletal problems that has required employees to seek active medical or orthopedic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the DASH index score | 12 months
  The DASH (Disability Arm, Shoulder, and Hand outcomes) is scored on a 0-100 scale. Higher score indicates greater disability. A change of 10 more points from baseline, noted at the end of the study will be considered significant
Change in ODI (Oswestry Disability Index) | 12 months
  The OSI is scored on a 0-100 scale, zero being with no disability and 100 with maximum disability possible. A change of 10 points from baseline will be considered significant

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Mankato, Mankato, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials